CLINICAL TRIAL: NCT06491797
Title: Booster of the "More Time for Patients" Program: a Cluster Randomized Controlled Trial
Brief Title: Booster of the "More Time for Patients" Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Thomas Agoritsas, Professor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PTPBooster
Record Dates: First submitted 2024-06-06; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Clinical Encounter Quality
Keywords: Health Care Quality, Access and Evaluation; Patient satisfaction; Job satisfaction; Inpatients; Pain Management
MeSH Terms: conditions — Patient Satisfaction; Agnosia

STUDY DESIGN:
Intervention Model Description: Intervention group will see immediate reactivation of the program where control intervention will be the program as it is usually applied before the application of the booster measure (applied delayed by three months).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate reactivation (Experimental): Our intervention will be booster measure of the existing PTP elements that will be designed for each unit that has been randomized to the immediate intervention group. The booster will consist in a reactivation through audit and feedback of 2-3 elements of the PTP program. The selection of the elements to boost will be done locally in each unit through a coordinated discussion between representants of the PTP organization and representants of the unit's medical and nursing professionals. This will create an adaptable intervention that will feature selected standards among the list of 36 existing standards. The boost will be performed over 3 months
  Interventions: Behavioral: Immediate reactivation
- Delayed reactivation (No Intervention): The control intervention will also be PTP as applied usually, in the control group before the application of the booster measure (applied delayed by three months).

INTERVENTIONS:
Behavioral: Immediate reactivation — Our intervention will be booster measure of the existing PTP elements that will be designed for each unit that has been randomized to the immediate intervention group. The booster will consist in a reactivation through audit and feedback of 2-3 elements of the PTP program. The selection of the elements to boost will be done locally in each unit through a coordinated discussion between representants of the PTP organization and representants of the unit's medical and nursing professionals. This will create an adaptable intervention that will feature selected standards among the list of 36 existing standards. The boost will be performed over 3 months
  Arms: Immediate reactivation

SUMMARY:
The goal of this clinical trial is to determine if reactivating a hospital program called "Plus de temps au service des patients" (PTP) can improve the quality of pain management for patients and increase job satisfaction among healthcare professionals. The main questions this study aims to answer are:

* Does reactivating PTP improve the quality of pain management?
* Does reactivating PTP increase healthcare professionals' job satisfaction? In this study, researchers will compare the effects of reactivating the program immediately to reactivating it after a 3-month delay.

Participants in the trial are healthcare professionals who will:

* Select 2 or 3 elements of the program they believe would be most beneficial to reactivate in their hospital units.
* Implement the selected elements for 3 months.
* Complete job satisfaction and burnout questionnaires before and after the study.

ELIGIBILITY:
Inclusion criteria for the units:

* Implementation of PTP finished at least 6 months previously
* Agreement to the study from both medical head of service and head of unit (IRES)

Inclusion criteria for healthcare professionals:

* Healthcare professionals >18 yo.
* Healthcare professionals working in a HUG service of medicine or surgery.
* Healthcare professionals include Physicians, Nurses, Assistant Nurses, Pharmacists, Physiotherapists and other physical therapists.
* Provided general informed consent.

Inclusion criteria for patients

* Patients hospitalised in one of the boosted units.
* Cognitive ability to provide satisfaction assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 764 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Timely delivery of appropriate analgesic | Timely is operationalized as maximum 6 hours before for reserve pain medication, and up to 1 hour after pain measurement for any medication appropriate to the level of pain.
  Quality of pain management as recorded through the timely delivery of an appropriate level painkiller after any pain Visual Analog Scale (VAS) ≥4. VAS score range from 0 to 10, 0 being no pain and 10 being the worse pain imaginable.

SECONDARY OUTCOMES:
Pain VAS documentation | 12 hours
  Patients stay will be divided in 12 hours segments and documentation will be considered adequate when 90% of the segments have at least 1 pain Visual Analog Scale score documented. VAS score range from 0 to 10, 0 being no pain and 10 being the worse pain imaginable.
Patient satisfaction - Picker | 1 week after discharge for every patients.
  Patient satisfaction is already routinely collected via continuous Picker satisfaction questionnaires. They are sent one week after patient discharge to all patients with a valid email address.
Patient satisfaction - daily | Every day from month 1 to month 3 corresponding to the period of study
  Daily patient satisfaction is already routinely collected in a 3 level scale going from 1 dissatisfied to 3 fully satisfied. Surveys are realized at the bedside, often by nurse assistant in the early afternoon.
Healthcare professionals' satisfaction | Once before the reactivation and once after (month 1 and month 3)
  Healthcare professionals' satisfaction will be evaluated using the satisfaction with work scale. All item range from extremely dissatisfied to extremely satisfied.
Healthcare professionals' burnout | Once before the reactivation and once after (month 1 and month 3)
  Burnout will be assessed using the Copenhagen burnout inventory. The Copenhagen Burnout Inventory is a three dimensions scale evaluating the personal, the professional and the relational components of burnout. Each dimension is scored on a scale ranging from 0 to 100, 0 being no burnout and 100 being the maximum burnout.
Healthcare professionals' risk of turnover | Once before the reactivation and once after (month 1 and month 3)
  Risk of turnover will be investigated by the following validated single item "If it were possible and you would keep a similar salary, would you like to change profession to take up another one or to keep the same profession but without patient care?" Three answers are possible: "No, I do not want to", "Perhaps", and "Yes, I do want to"
Healthcare professional's absenteeism rate | At month 1, 2 and 3 corresponding to the period of study
  If given consent by the participants, individual monthly absenteeism rate will be extracted from the human resources of the hospital. For all others, absenteeism rate will be extracted aggergated at the unit level.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Agoritsas, MD, PhD, Principal Investigator — University Hospital, Geneva; Delphine S. Courvoisier, PhD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buclin CP, Burgisser N, Mongin D, Le Mauguen A, Farhoumand PD, Berner A, Daverio JE, Barrios J, Reny JL, Courvoisier DS, Agoritsas T. Impact of a booster intervention of the 'More Time at Patients' Side' programme on patients and healthcare professionals in a Swiss hospital: protocol for a cluster randomised controlled trial. BMJ Open. 2026 Jan 13;16(1):e104027. doi: 10.1136/bmjopen-2025-104027. PMID 41529885